CLINICAL TRIAL: NCT02223052
Title: A Phase 1, Open-label, Multicenter, Randomized, 2-Period, Crossover Study to Evaluate the Bioequivalence and Food Effect Bioavailability of CC-486 (Oral Azacitidine) Tablets in Adult Cancer Subjects
Brief Title: Bioequivalence & Food Effect Study in Patients With Solid Tumor or Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-486-CAGEN-001
Expanded Access: NCT03723135 (Approved for marketing)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Hematological Neoplasms; Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Lymphoma; Multiple Myeloma; Acute Myeloid Leukemia; Leukemia; Myelodysplastic Syndromes; Neoplasms; Melanoma; Breast Cancer; Metastatic Breast Cancer; Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Renal Cell Carcinoma; Glioblastoma Multiforme; Osteosarcoma; Sarcoma; Thyroid Cancer; Genitourinary
Keywords: CC-486; Oral Azacitidine; Soli Tumor Malignancy; Hematological Malignancy; Leukemia; Lymphoma; Multiple Myeloma; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Neoplasms; Melanoma; Breast Cancer; Metastatic Breast Cancer; Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Renal Cell Carcinoma; Glioblastoma Multiforme; Brain Cancer; Kidney Cancer; Lung cancer; Blood Cancer; Thyroid Cancer; Bone Cancer; Bone Metastasis; Testicular Cancer; Prostate Cancer; Bladder Cancer; Ovarian Cancer; Skin Cancer; Cancer general; Survival; Chemotherapy; Targeted Therapy; Genitourinary; MM; MDS; AML; NHL; HL; MBC; NSCLC; SCLC; GBM
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma; Multiple Myeloma; Leukemia, Myeloid, Acute; Leukemia; Myelodysplastic Syndromes; Neoplasms; Melanoma; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Glioblastoma; Osteosarcoma; Sarcoma; Thyroid Neoplasms; Brain Neoplasms; Kidney Neoplasms; Lung Neoplasms; Bone Neoplasms; Testicular Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Skin Neoplasms | interventions — cc-486; Azacitidine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CC-486 Arm 1 (Oral Azacitidine) Dosing Sequence 1 (Experimental): Two 150-mg tablets of CC-486 under fasting condition on PK dosing Day 1, followed by one 300-mg tablet of CC-486 on PK dosing Day 2; If PI chooses to treat the patient in the extension phase with Azacitidine, Vidaza (Azacitidine for Injection) 75 mg/m2 intravenously (IV) or subcutaneously (SC) daily x 7 days every 4 weeks for less than or equal to 6 (28-day) cycles will be administered.
  Interventions: Drug: CC-486; Drug: Vidaza
- CC-486 Arm 2 (Oral Azacitidine) Dosing Sequence 1 (Experimental): One 300-mg tablet of oral CC-486 under fasting condition on PK dosing Day 1, followed by one 300-mg tablet of oral CC-486 under fed condition on PK dosing Day 2; If PI chooses to treat the patient in the extension phase with Azacitidine, Vidaza (Azacitidine for Injection) 75 mg/m2 intravenously (IV) or subcutaneously (SC) daily x 7 days every 4 weeks for less than or equal to 6 (28-day) cycles will be administered.
  Interventions: Drug: CC-486; Drug: Vidaza
- CC-486 Arm 1 (Oral Azacitidine) Dosing Sequence 2 (Experimental): One 300-mg tablets of CC-486 under fasting condition on PK dosing Day 1, followed by two 150-mg tablets on PK dosing Day 2; If PI chooses to treat the patient in the extension phase with Azacitidine, Vidaza (Azacitidine for Injection) 75 mg/m2 intravenously (IV) or subcutaneously (SC) daily x 7 days every 4 weeks for less than or equal to 6 (28-day) cycles will be administered.
  Interventions: Drug: CC-486; Drug: Vidaza
- CC-486 Arm 2 (Oral Azacitidine) Dosing Sequence 2 (Experimental): One 300-mg tablet of oral CC-486 under fed condition on PK dosing Day 1, followed by one tablet of 300-mg oral CC-486 under fasted conditions on PK dosing Day 2; if PI chooses to treat the patient in the extension phase with Azacitidine, Vidaza (Azacitidine of Injection) 75 mg/m2 intravenously (IV) or subcutaneously (SC) daily x 7 days every 4 weeks for less than or equal to 6 (28-day) cycles will be administered.
  Interventions: Drug: CC-486; Drug: Vidaza

INTERVENTIONS:
Drug: CC-486 — Arm 1: Two 150-mg tablets of CC-486 on Day 1 and 1 x 300 mg CC-486 on Day 2 Arm 2: 1 x 300mg tablet of CC 486 on Day 1 and 2 x 150mg CC-486 on Day 2
  Other Names: Oral Azacitdine
Drug: Vidaza — 75mg/m^2 IV or SC daily x 7 days every 4 weeks for ≤ 6 (four-week) cycles
  Other Names: Azacitidine for Injection; AZA

SUMMARY:
This is a Phase 1, open-label, multicenter, randomized, 2-stage crossover study consisting of 2 phases:

Stage I - Pharmacokinetics (Bioequivalence), with an Extension Stage II - Pharmacokinetics (Food Effect) with an Extension

This study will enroll approximately 60 subjects in stage I and 60 subjects in stage II with hematologic or solid tumor malignancies, excluding gastrointestinal tumors and tumors that have originated or metastasized to the liver for which no standard treatment exists or have progressed or recurred following prior therapy. Subjects must not be eligible for therapy of higher curative potential where an alternative treatment has been shown to prolong survival in an analogous population. Approximately 23 sites in the US and 2 in Canada will participate in this study.

DETAILED DESCRIPTION:
Stage I - Pharmacokinetics (Bioequivalence)

Subjects will be randomized to receive CC-486 300 mg orally on each of the two pharmacokinetic (PK) study days based on the dosing sequences they are randomized to:

Dosing Sequence 1: 2x150 mg tablets followed by 1x30 mg tablet. Dosing Sequence 2: 1x300 mg tablet followed by 2x150 mg tablets. Each dose will be administered in the clinic at least 48 hours apart between PK dosing day 1 and PK dosing day 2 over a period no longer than 10 days under fasted conditions.

Stage II - Pharmacokinetics (Food Effect)

Subjects will be randomized to receive CC-486 300 mg orally on each of the two PK study days based on the dosing sequences they are randomized to:

Dosing Sequence 1: 1x300 mg tablet under fasted condition followed by 1x300 mg tablet under fed condition.

Dosing Sequence 2: 1x300 mg tablet under fed condition followed by 1x300 mg tablet under fasted condition.

Each dose will be administered in the clinic at least 48 hours apart between PK dosing day 1 and PK dosing day 2 over a period no longer than 10 days. The sponsor will generate the randomization scheme and assign subjects upon enrollment to the appropriate sequence for dosing:

Fasted condition: following an overnight fast of at least 10 hours, subjects will ingest oral Azacitidine with 240 mL of room temperature water. Subjects must fast for a minimum of 4 hours following oral Azacitidine administration. Subjects may drink water as desired, except for 1 hour before and 1 hour after oral Azacitidine administration.

Fed condition: following an overnight fast of at least 10 hours and following the performance of all required pre-dose assessments, subjects randomized to receive test medication in a fed state will begin ingesting a breakfast meal 30 (±5) minutes prior to the planned administration of oral Azacitidine. They will continue the entire meal within 20 to 25 minutes (no less than 20 minutes) from the time the meal is served. Subjects will then ingest oral Azacitidine with 240 mL of room temperature water. Subjects must fast a minimum of 4 hours following oral Azacitidine administration. Subjects may drink water as desired, except for 1 hour before and 1 hour after administration of oral Azacitidine.

Extension Phase (for subjects who have completed PK Stage I or Stage II) Subjects continuing beyond the pharmacokinetics phase (Stage I or Stage II) will enter the extension phase of the study at the discretion of the investigator to receive < 6 (four-week) cycles of Vidaza 75 mg/m2 IV or SC daily for 7 days in the clinic and repeat every 4 weeks per prescribed label at the discretion of the investigator for ≤ 6 (four-week) cycles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  1. Age ≥ 18 years of age at the time of signing the informed consent document.
  2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
  3. Documented diagnosis of any of the following:

     1. Myelodysplastic Syndrome (MDS) according to the World Health Organization (WHO) 2008 classification
     2. Acute myeloid leukemia (AML)
     3. Multiple myeloma (MM), limited to those patients for whom standard curative or palliative treatments do not exist or are no longer effective
     4. Non-Hodgkin's lymphoma (NHL), limited to those patients for whom standard curative or palliative treatment do not exist or are no longer effective,
     5. Hodgkin's lymphoma (HL), limited to those patients for whom standard curative or palliative treatment do not exist or are no longer effective
     6. Metastatic or inoperable solid tumors* (except gastrointestinal tumors or tumors that originated or metastasized to the liver) for which no standard treatment exists, or have progressed or recurred following prior therapy.

        * Subjects must not be eligible for therapy of higher curative potential where an alternative treatment has been shown to prolong survival in an analogous population.
  4. Patients with a history of treated brain metastases should be clinically stable for ≥ 4 weeks prior to signing the informed consent. Glucocorticoid therapy for central nervous system (CNS) edema is permitted if ≤ 20 mg of prednisolone (or equivalent).
  5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
  6. Have a life expectancy of ≥ 3 months.
  7. Have stable renal function without dialysis for at least 2 months prior to Investigational Product (IP) administration defined by:

     1. Serum creatinine < 2.5 x the upper limit of normal (ULN)
     2. An average calculated creatinine clearance > 30 mL/min/1.73 m^2
  8. Have organ and marrow function at the screening and pre-dose visits as defined by:

     1. Hemoglobin ≥ 8 g/dL
     2. Absolute neutrophil count (ANC) ≥ 0.75 x 10^3/uL without treatment with a myeloid growth factor within 3 days prior to first dose of IP
     3. Platelets ≥ 30 x 10^3/uL
     4. Total bilirubin ≤ 1.5 x Upper Limits of Normal (ULN)
     5. Aspartate aminotransferase (AST) ≤ 2 x ULN
     6. Alanine aminotransferase (ALT) ≤ 2 x ULN
  9. Have a 12-lead Electrocardiogram (ECG) that is not clinically significant at screening, as determined by the investigator
  10. Females of childbearing potential (FCBP) may participate, providing the subject meets the following conditions:

      * Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) or agree to practice true abstinence throughout the study, and for 3 months following the last dose of IP; and
      * Negative serum pregnancy test at screening (sensitivity of at least 25 mIU/mL); (Note that the screening serum pregnancy test can be used as the test prior to starting IP in the pharmacokinetics phase if it is performed within the 72-hour timeframe), and
      * Negative serum or urine pregnancy test (investigator's discretion; sensitivity of at least 25 mIU/mL) within 72 hours prior to starting IP in the extension phase. (Note: subjects must have negative serum or urine pregnancy test prior to dosing on Day 1 of each treatment cycle in the extension phase.)
  11. Male subjects must:

      a. Practice true abstinence* or agree to the use of at least two physician-approved contraceptive methods throughout the course of the study and should avoid fathering a child during the course of the study for at least 3 months following the last dose of IP.

      * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
  12. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Women who are pregnant or nursing (lactating).
2. Gastrointestinal tumors, tumors that have originated or metastasized to the liver, or other tumors known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
3. Had chemotherapy or radiotherapy within 4 weeks prior to the first day of Investigational Product (IP) administration.
4. Have been treated with an investigational agent within 4 weeks prior to the first day of IP administration.
5. Have ongoing clinically significant adverse event(s) due to prior treatments administered as determined by the investigator.
6. Significant active cardiac disease within the previous 6 months, including:

   * New York Heart Association (NYHA) class IV congestive heart failure
   * Significant cardiac arrhythmia or unstable angina or angina requiring surgical or medical intervention; and/or
   * Myocardial infarction
7. Have known or suspected hypersensitivity to azacitidine or any other ingredient used in the manufacturing of Azacitidine.
8. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
9. History of inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis), celiac disease, prior gastrectomy, gastric bypass, upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption of the study drug and/or predispose the subject to an increased risk of gastrointestinal toxicity.
10. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
11. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
12. Any condition that confounds the ability to interpret data from the study
13. Impaired ability to swallow oral medication
14. Any condition that confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Cmax - Stage I (Bioequivalence) | Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose
  The observed maximum concentration
Pharmacokinetics Tmax - Stage I (Bioequivalence) | Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose
  The observed time to first maximum concentration
Pharmacokinetics AUC-t - Stage I (Bioequivalence) | Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose
  Area under the concentration-time curve from time zero to the last quantifiable time point calculated by the linear trapezoidal rule
Pharmacokinetics AUC-infinity - Stage I (Bioequivalence) | Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose
  Area under the concentration time-curve from time zero to infinity, calculated by the linear trapezoidal rule and extrapolated to infinity. It will be calculated as AUC∞ = [AUCt + Ct/λz]. Ct is the last quantifiable concentration
Pharmacokinetics λz (Terminal Rate) - Stage I (Bioequivalence) | Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.3.5, 4, 6, and 8 hours post-dose
  Terminal phase rate constant, determined by linear regression of the terminal points of the log-linear concentration-time curve
Pharmacokinetics Terminal Half-Life (t½) - Stage I (Bioequivalence) | Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose
  Terminal phase half-life, calculated according to the following equation: t½ = 0.693/λz
Pharmacokinetics Apparent total clearance (CL/F) - Stage I (Bioequivalence) | Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose
  Apparent total clearance, calculated as Dose/AUC∞
Pharmacokinetics Apparent volume of distribution (Vd/F) - Stage I (Bioequivalence) | Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose
  Apparent volume of distribution, calculated according to the equation: Vd/F = (CL/F) / λz
Pharmacokinetics Cmax - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  The observed maximum concentration
Pharmacokinetics Tmax - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  The observed time to first maximum concentration
Pharmacokinetics AUC-t - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  Area under the concentration-time curve from time zero to the last quantifiable time point calculated by the linear trapezoidal rule.
Pharmacokinetics AUC-infinity - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  Area under the concentration time-curve from time zero to infinity, calculated by the linear trapezoidal rule and extrapolated to infinity. It will be calculated as AUC∞ = [AUCt + Ct/λz]. Ct is the last quantifiable concentration.
Pharmacokinetics λz (Terminal Rate) - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  Terminal phase rate constant, determined by linear regression of the terminal points of the log-linear concentration-time curve
Pharmacokinetics Terminal Half-Life (t½) - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  Terminal phase half-life, calculated according to the following equation: t½ = 0.693/λz
Pharmacokinetics Apparent total clearance (CL/F) - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  Apparent total clearance, calculated as Dose/AUC∞
Pharmacokinetics Apparent volume of distribution (Vd/F) - Stage II (Food Effect Bioavailability) | PK Dosing Day 1 and PK Dosing Day 2 prior to each dose administration of IP (CC-486), known as pre-dose, and over the 8-hour period following each dose administration of IP (CC-486) at 0.25, 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 6, and 8 hours post-dose.
  Apparent volume of distribution, calculated according to the equation: Vd/F = (CL/F) / λz

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 18 months
  Adverse Event (AE) is defined as any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Du Lam, MD, Study Director — Celgene
Locations (10):
- United States (10):
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of Iowa, Iowa City, Iowa
  - Henry Ford Health System, Detroit, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Greenville Hospital System, Greenville, South Carolina
  - Vanderbilt- Ingram Cancer Center, Nashville, Tennessee
  - The Methodist Hospital Research Institute l, Houston, Texas